CLINICAL TRIAL: NCT07272408
Title: Impact of Remote Ischemic Conditioning in Patients Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Remote Ischemic Conditioning in Patients Undergoing Primary Percutaneous Coronary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Ahmed Yousry Mousa, Resident of Cardiology, Helwan University, Helwan, Egypt, Helwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 40-2022
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Remote; Ischemic Conditioning; Primary Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote ischemic conditioning (Experimental): Remote ischemic conditioning (RIC) was applied to those patients.
  Interventions: Procedure: Remote ischemic conditioning
- Normal primary percutaneous coronary intervention (Active Comparator): Patients followed the standard primary percutaneous coronary intervention pathway.
  Interventions: Procedure: Normal primary percutaneous coronary intervention

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Remote ischemic conditioning (RIC) was applied to those patients.
  Arms: Remote ischemic conditioning
Procedure: Normal primary percutaneous coronary intervention — Patients followed the standard primary percutaneous coronary intervention pathway.
  Arms: Normal primary percutaneous coronary intervention

SUMMARY:
This study aimed to detect the effects of remote ischemic conditioning on infarct size, global contractility, morbidity, mortality, and renal function in patients undergoing primary percutaneous coronary intervention.

DETAILED DESCRIPTION:
Myocardial infarction (MI) generally refers to segmental (regional) myocardial necrosis, typically endocardial in location, secondary to occlusion of an epicardial artery.

Primary percutaneous coronary intervention (PPCI) is a reperfusion therapy that is carried out in patients who usually have ST-segment elevation MI (STEMI) within a specific time window.

During ischemia, metabolic acidosis occurs due to anaerobic metabolism, and ischemic injury ensues. After restoration of blood supply, reactive oxygen species (ROS) production and local inflammation increase secondary injury.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 and less than 75 years old.
* Both sexes.
* Patients with new ST-segment elevation at the J-point in V1:V6 leads with the cut-point: ≥ 1mm other than leads V2-V3 where the following cut-points apply: ≥ 2mm in men ≥ 40 years; ≥ 2.5mm in men < 40 years, or ≥ 1.5mm in women regardless of age.
* Patients with new left bundle branch block (LBBB).

Exclusion Criteria:

* ST-segment elevation myocardial infarction (STEMI) with cardiogenic shock.
* Severe comorbidities (uncontrolled hypertension, morbid obesity, recent cerebrovascular stroke, respiratory failure, sepsis, and stage 4 & 5 malignancy).
* End-stage renal disease on hemodialysis.
* Previous coronary artery bypass graft surgery (CABG).
* Myocardial infarct within the previous 30 days.
* Multi-vessel coronary artery disease.
* Failure of culprit vessel recanalization.
* Conditions precluding use of remote conditioning ie: paresis of upper limb.
* Life expectancy of less than 1 year due to a non-cardiac pathology.
* Patients who receive nephrotoxic drugs such as non-steroidal anti-inflammatory drugs and aminoglycosides.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Cardiac death | 1 month post-procedure
  Incidence of cardiac death was recorded.

SECONDARY OUTCOMES:
Hospitalization for heart failure | 1 month post-procedure
  Hospitalization for heart failure post-randomization in the intention-to-treat population was assessed.
Contrast induced nephropathy | 1 month post-procedure
  Contrast induced nephropathy was assessed.
Incidence of adverse events | 1 month post-procedure
  Incidence of adverse events was recorded.
Renal impairment | 1 month post-procedure
  Renal impairment was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Helwan University, Helwan, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.